CLINICAL TRIAL: NCT04276675
Title: Cardiac Rehabilitation Programme in Patients Following Hospitalisation for Decompensated Chronic Heart Failure: the Development of an Intervention to Improve Patient Acceptance of Referral.
Brief Title: CR: Developing an Intervention to Improve Acceptance of Referral in HF
Acronym: CREATE-HF
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0739
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure; Frailty
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: There are proven benefits to people with chronic heart failure (CHF) participating in a cardiac rehabilitation (CR) programme, however uptake remains disappointingly low. Admission to hospital presents a significant opportunity to offer CR referral to such a patient population. It is believed that up to 75% of patients with CHF show signs of frailty at discharge which might impact on the rate of patients' acceptance of referral to CR.

Aim: To explore the impact of frailty on patient acceptance of referral to CR following admission to hospital with an episode of decompensated CHF.

Methods and expected outcome: We will conduct an observational study assessing the relationship between frailty and acceptance of referral to CR in this patient population. It will also explore what factors impact that relationship including demographic factors, measures of self-care and patient activation measure (PAM).

DETAILED DESCRIPTION:
Trial Design: Mixed method approach to development of an intervention: observational cohort study, semi-structured interviews, focus groups, staff survey, theory informed intervention development using 'The Behaviour Change Wheel'.

Trial Participants:

1. Patients admitted to hospital for an episode of decompensated heart failure who have been referred to the Heart Failure Nursing Service (HFNS) and are eligible for referral for cardiac rehabilitation.
2. Patients who have been referred to cardiac rehabilitation from the HFNS, Cardiology outpatients and general practice.
3. Health care professionals involved in the referral to or provision of cardiac rehabilitation services for people with chronic heart failure

Planned Sample Size:

203 patients in observational study; 8 to 40 participants in semi-structured interviews;10 to 15 health care professionals in focus groups; 40 health care professionals questionnaire

Follow-up duration:

Part 1 of the study: Observational Cohort: from discharge to 6 weeks post discharge; Part 2 of the study: Semi-structured interviews: participants have single semi-structured interview and given the opportunity to feedback on final proposed intervention Focus groups: cardiac rehabilitation team health care professionals participate in one focus group and feedback on final proposed intervention. Part 3 of study: Health care professional: single participation in survey and subgroup of HCP feedback on final proposed intervention

Planned Trial Period 24 months (including feasibility study of intervention)

Primary Objective: The primary objective of this study is to determine the key modifiable patient related factors associated with the acceptance of referral to cardiac rehabilitation in patients post discharge following an episode of decompensated chronic heart failure.

Secondary Objectives: Using the Behaviour Change wheel synthesize the data from the observational study, stakeholder perspectives and the literature on behaviour change interventions, develop a theory based intervention to increase the uptake of referral to cardiac rehabilitation in patients post discharge following an episode of decompensated chronic heart failure.

Primary Endpoint:

Observational study: Uptake of referral to cardiac rehabilitation by patients following an episode of decompensated heart failure at baseline visit.

Semi-structured interviews, focus groups and staff survey: Identify patient, and health care professional perceived barriers and facilitators to the uptake of referral to cardiac rehabilitation by patients following an episode of decompensated heart failure.

Secondary Endpoints:

Observational study: Uptake of referral to cardiac rehabilitation by patients following an episode of decompensated heart failure at 6 weeks post discharge.

Semi-structured interviews, focus groups and staff survey: Identify the impact of COVID 19 pandemic on the uptake of referral and participation in cardiac rehabilitation by patients following an episode of decompensated heart failure.

In consultation with experts in theory based interventions, data from all steps of the programme of study will be used to develop an intervention aimed at improving rate of acceptance of referral to CR in this patient population.

Further stakeholder involvement The intervention will be presented back in written form to interviewees and focus group members for further comment either written or via telephone contact. Health care professionals (HFNS team and CR team) will be invited for feedback on expected effectiveness and acceptability following which further adaptation of the intervention may occur

ELIGIBILITY:
Observational study:

Inclusion Criteria:

* Clinical diagnosis of chronic heart failure confirmed by cardiac imaging.
* Current admission for which the primary reason was decompensated heart failure requiring IV diuretics
* Referred to the acute trusts heart failure nursing service
* Able to give informed consent
* Able to communicate in spoken English

Exclusion Criteria:

* Contraindications to participating in cardiac rehabilitation as detailed in ESC consensus statement e.g. uncontrolled hypertension severe aortic stenosis, unstable angina
* Moderate to severe cognitive impairment
* Patients with severe dependence prior to index admission (inability to carry out ADL)
* Admitted from a nursing home
* Resident 'out of area'
* Significant co-morbidities that would limit participation in a cardiac rehabilitation programme e.g. neurodegenerative conditions
* Previous recruitment onto this study

Semi-structured interviews: Purposive sampling

Inclusion criteria:

* Patients with chronic heart failure who fulfil the criteria for referral to the cardiac rehabilitation service will be eligible to participate in the interviews if they are:
* Age 18 years or over
* Have a clinical diagnosis of CHF confirmed by cardiac imaging.
* Referred to the acute trusts heart failure nursing service and/or cardiac rehabilitation team
* Able to give informed consent
* Able to communicate in spoken English

Exclusion criteria:

* Contraindications to participating in cardiac rehabilitation as detailed in ESC consensus statement (See Appendix D) e.g. uncontrolled hypertension, severe aortic stenosis, unstable angina
* Moderate to severe cognitive impairment
* Nursing home resident
* Significant co-morbidities that would limit participation in a cardiac rehabilitation programme e.g. neurodegenerative conditions
* Previous recruitment onto this study

Focus groups: convenience sampling

Inclusion criteria:

Staff from study site who are involved in the provision of cardiac rehabilitation to people with heart failure will be eligible to participate in the focus group.

Survey: convenience sampling

Inclusion criteria:

Health care professionals who refer to or deliver cardiac rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational cohort: All patients admitted to the participating hospital with an episode of decompensated chronic heart failure and referred to the Heart Failure Nursing Service (HFNS) who are eligible for referral to cardiac rehabilitation.
  Semi-structured interviews: Participants of observational study; people with heart failure eligible for CR and referred to either the acute trust's heart failure nursing service and/ or cardiac rehabilitation team.
  Survey: Health care professionals involved in delivering or referring to cardiac rehabilitation to people with chronic heart failure.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Acceptance of referral to cardiac rehabilitation | Within 7 days from baseline visit
  Identify whether participant has been referred to CR
Qualitative evaluation of impact of offer of referral to cardiac rehabilitation service | 6 weeks
  Health care professionals offer referral to cardiac rehabilitation to people with heart failure as part of their ongoing treatment. Interviews and focus groups will be used to identify patient and health care professional perceived barriers and facilitators to the uptake of referral to cardiac rehabilitation by patients. Outcome measures from these cannot be counted and the data will be analysed using qualitative methods to identify themes representing the meanings associated with the participants' disclosures.

SECONDARY OUTCOMES:
Acceptance of referral to cardiac rehabilitation | 6 weeks post discharge
  Identify whether participant has been referred to CR
Qualitative evaluation of impact of COVID 19 on acceptance of referral to cardiac rehabilitation service | 6 weeks
  This study was recruiting during the COVID 19 pandemic. Interviews and focus groups will be used to identify the impact of COVID 19 on the uptake of referral to cardiac rehabilitation by people with heart failure. Outcome measures from these cannot be counted and data will be analysed using qualitative methods to identify themes representing meanings associated with participants' disclosures.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Waterhouse, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided